CLINICAL TRIAL: NCT05893472
Title: The Second Affiliated Hospital of Kunming Medical University
Brief Title: A Study on the Efficacy and Safety of Venetoclax Combined With HAA Regimen in Newly Diagnosed Young AML.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZePing Zhou (Other)
Collaborators: Handan Central Hospital (Other); Taian City Central Hospital (Other); Tianjin People's Hospital (Other); Guizhou Provincial People's Hospital (Other); Second Xiangya Hospital of Central South University (Other); Western War Zone General Hospital (Unknown)
Responsible Party: Sponsor-Investigator, ZePing Zhou, Dr., The Second Affiliated Hospital of Kunming Medical University
Organization: The Second Affiliated Hospital of Kunming Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEN-PJ-KE-2023-125
Record Dates: First submitted 2023-04-24; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukemia; Venetoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The treatment group receiving the combination of venetoclax and HAA regimen. (Experimental): Received induction therapy protocol： Docetaxel (HHT) 2.5mg/㎡/day, days 3-7 Aclarubicin (Acla) 20mg/day, days 3-7 Cytarabine (Ara-c) 100mg/㎡/day, days 3-7 (given as a 24-hour infusion) Venetoclax (VEN): 100mg on day 1, 200mg on day 2, and 400mg on days 3-8.
  Interventions: Combination Product: combination of venetoclax and HAA regimen

INTERVENTIONS:
Combination Product: combination of venetoclax and HAA regimen — Using the combination of venetoclax and HAA regimen as induction therapy in young, newly diagnosed adult acute myeloid leukemia patients under the age of 60.

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of the combination of venetoclax and HAA regimen in young, newly diagnosed acute myeloid leukemia patients under the age of 60.

ELIGIBILITY:
Inclusion Criteria:

* The eligible subjects for enrollment in this study must meet all of the following criteria:

  1. Patients with acute myeloid leukemia (excluding APL) who meet the diagnostic criteria of the World Health Organization (WHO) 2016 classification.
  2. Patients with AML and multilineage dysplasia (MDS) and/or myeloproliferative neoplasms (MPN) who meet the WHO criteria without prior history of MDS or MPN.
  3. Patients with AML who are not classified separately according to the WHO classification, except for those with acute megakaryoblastic leukemia with bone marrow fibrosis or myeloid sarcoma.
  4. Age greater than 16 years and less than 60 years, regardless of gender.
  5. Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0-2.
  6. Requirements for laboratory parameters (within 7 days prior to treatment initiation) include: aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤3 times the upper limit of normal (ULN); serum bilirubin ≤2×ULN; serum cardiac enzyme <2.0×ULN; serum creatinine ≤2.0×ULN; and echocardiogram (ECHO)-determined ejection fraction within the normal range.
  7. A signed informed consent form is required before any study-specific procedures are performed. Patients 18 years and older may sign the informed consent form themselves or have it signed by their next of kin. Patients under 18 years of age must have the informed consent form signed by their legal guardian. In consideration of the patient's medical condition, if it is not in the patient's best interest to sign the form, the legal guardian or patient's next of kin may sign the form on the patient's behalf.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from this study:

  1. Previously treated patients (including those who have undergone induction chemotherapy regardless of treatment response).
  2. Secondary leukemia (including therapy-related AML subtype according to the World Health Organization (WHO) classification and those with a history of MDS and/or MPD).
  3. Concomitant hematologic diseases (such as hemophilia or myelofibrosis) deemed unsuitable for inclusion by the investigator; individuals with prior abnormal blood counts are allowed to participate if they have been previously excluded from MDS and MPD.
  4. Other malignant tumors requiring treatment.
  5. Pregnant or lactating women. Female participants of childbearing potential must have a negative pregnancy test within 7 days prior to the start of the trial. Male or female participants must take contraceptive measures during the trial and for 3 years after completion of treatment.
  6. Significant abnormalities in liver or kidney function beyond the inclusion criteria.
  7. Active heart disease, defined as one or more of the following:

  <!-- -->

  1. History of uncontrolled or symptomatic angina pectoris;
  2. Myocardial infarction within 6 months prior to enrollment;
  3. History of arrhythmia requiring medication or with severe clinical symptoms;
  4. Uncontrolled or symptomatic congestive heart failure (> NYHA class 2);
  5. Ejection fraction below the lower limit of the normal range. 8. Severe infectious diseases (e.g., unhealed tuberculosis or pulmonary aspergillosis).

  9. Participants deemed unsuitable for inclusion by the investigator.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 12 months
  which evaluates the efficacy of patient induction therapy, including complete remission (CR), complete remission with incomplete blood count recovery (CRi), and morphologic leukemia-free state (MLFS)

SECONDARY OUTCOMES:
Minimal residual disease (MRD) | up to 12 months
  MRD percentage
overall survival (OS) | up to 12 months
  Overall Survival (OS) is used to evaluate all patients enrolled in a clinical trial, from the date of enrollment until death from any cause or the date of last follow-up for surviving patients.
relapse-free survival (RFS) | up to 12 months
  Relapse-Free Survival (RFS) is only used to evaluate patients who achieve complete remission (CR) through reinduction therapy. RFS is defined as the time from achievement of CR until death from any cause, relapse, or the date of last follow-up.
30-day mortality rate | Within 30 days after starting the medication
  The 30-day mortality rate is used to evaluate all patients enrolled in a clinical trial, and is defined as the percentage of patients who die within 30 days of starting chemotherapy.
adverse drug reactions | up to 12 months
  Adverse drug reactions during chemotherapy and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: DanQi Deng, Study Chair — The Second Affiliated Hospital, Kunming Medical University
Locations (1):
- The Second Affiliated Hospital of Kunming Medical University., Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Del Poeta G, Venditti A, Del Principe MI, Maurillo L, Buccisano F, Tamburini A, Cox MC, Franchi A, Bruno A, Mazzone C, Panetta P, Suppo G, Masi M, Amadori S. Amount of spontaneous apoptosis detected by Bax/Bcl-2 ratio predicts outcome in acute myeloid leukemia (AML). Blood. 2003 Mar 15;101(6):2125-31. doi: 10.1182/blood-2002-06-1714. Epub 2002 Nov 7. PMID 12424199
- [Background] Mei M, Aldoss I, Marcucci G, Pullarkat V. Hypomethylating agents in combination with venetoclax for acute myeloid leukemia: Update on clinical trial data and practical considerations for use. Am J Hematol. 2019 Mar;94(3):358-362. doi: 10.1002/ajh.25369. Epub 2018 Dec 13. PMID 30499168
- [Background] DiNardo CD, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Wei AH, Konopleva M, Dohner H, Letai A, Fenaux P, Koller E, Havelange V, Leber B, Esteve J, Wang J, Pejsa V, Hajek R, Porkka K, Illes A, Lavie D, Lemoli RM, Yamamoto K, Yoon SS, Jang JH, Yeh SP, Turgut M, Hong WJ, Zhou Y, Potluri J, Pratz KW. Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia. N Engl J Med. 2020 Aug 13;383(7):617-629. doi: 10.1056/NEJMoa2012971. PMID 32786187
- [Background] Wei AH, Strickland SA Jr, Hou JZ, Fiedler W, Lin TL, Walter RB, Enjeti A, Tiong IS, Savona M, Lee S, Chyla B, Popovic R, Salem AH, Agarwal S, Xu T, Fakouhi KM, Humerickhouse R, Hong WJ, Hayslip J, Roboz GJ. Venetoclax Combined With Low-Dose Cytarabine for Previously Untreated Patients With Acute Myeloid Leukemia: Results From a Phase Ib/II Study. J Clin Oncol. 2019 May 20;37(15):1277-1284. doi: 10.1200/JCO.18.01600. Epub 2019 Mar 20. PMID 30892988
- [Background] DiNardo CD, Maiti A, Rausch CR, Pemmaraju N, Naqvi K, Daver NG, Kadia TM, Borthakur G, Ohanian M, Alvarado Y, Issa GC, Montalban-Bravo G, Short NJ, Yilmaz M, Bose P, Jabbour EJ, Takahashi K, Burger JA, Garcia-Manero G, Jain N, Kornblau SM, Thompson PA, Estrov Z, Masarova L, Sasaki K, Verstovsek S, Ferrajoli A, Weirda WG, Wang SA, Konoplev S, Chen Z, Pierce SA, Ning J, Qiao W, Ravandi F, Andreeff M, Welch JS, Kantarjian HM, Konopleva MY. 10-day decitabine with venetoclax for newly diagnosed intensive chemotherapy ineligible, and relapsed or refractory acute myeloid leukaemia: a single-centre, phase 2 trial. Lancet Haematol. 2020 Oct;7(10):e724-e736. doi: 10.1016/S2352-3026(20)30210-6. Epub 2020 Sep 5. PMID 32896301
- [Background] DiNardo CD, Lachowiez CA, Takahashi K, Loghavi S, Xiao L, Kadia T, Daver N, Adeoti M, Short NJ, Sasaki K, Wang S, Borthakur G, Issa G, Maiti A, Alvarado Y, Pemmaraju N, Montalban Bravo G, Masarova L, Yilmaz M, Jain N, Andreeff M, Jabbour E, Garcia-Manero G, Kornblau S, Ravandi F, Konopleva MY, Kantarjian HM. Venetoclax Combined With FLAG-IDA Induction and Consolidation in Newly Diagnosed and Relapsed or Refractory Acute Myeloid Leukemia. J Clin Oncol. 2021 Sep 1;39(25):2768-2778. doi: 10.1200/JCO.20.03736. Epub 2021 May 27. PMID 34043428
- [Background] Jin J, Wang JX, Chen FF, Wu DP, Hu J, Zhou JF, Hu JD, Wang JM, Li JY, Huang XJ, Ma J, Ji CY, Xu XP, Yu K, Ren HY, Zhou YH, Tong Y, Lou YJ, Ni WM, Tong HY, Wang HF, Mi YC, Du X, Chen BA, Shen Y, Chen Z, Chen SJ. Homoharringtonine-based induction regimens for patients with de-novo acute myeloid leukaemia: a multicentre, open-label, randomised, controlled phase 3 trial. Lancet Oncol. 2013 Jun;14(7):599-608. doi: 10.1016/S1470-2045(13)70152-9. Epub 2013 May 9. PMID 23664707